CLINICAL TRIAL: NCT04767334
Title: The Effect of Lower Body Positive Pressure Treadmill Training on Postural Control and Gait Function in Individuals With Chronic Stroke
Brief Title: The Effect of Lower Body Positive Pressure Treadmill Training on Individuals With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Sattam Almutairi, Assistant professor, Qassim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-05-04
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gait training on Lower body positive pressure (Experimental): All participants will have gait training for 40 minutes a day, for three days a week, for six weeks. On session one, the lower body positive pressure chamber will be set to unload 50% of patient's body weight.On the following sessions, the percentage of unload patient's body weight will be decrease depends on the patient's comfort.
  The physical therapist assistance and treadmill speed will be evaluated and altered based on the patient's capacity. The participants can take a rest whenever his/her need during walking. The rest time will be measured and documented.
  Interventions: Device: Anti-Gravity Treadmill

INTERVENTIONS:
Device: Anti-Gravity Treadmill — Each participant will started with a 5 - 10 minute warm-up on a standard cycle ergometer, manual and therapeutic therapy for upper extremity, and gait training using LBPP. Manual and therapeutic therapy will consist of passive and active ROM, joint mobilization, passive and active stretch, manual resistance exercise, and activities of daily life (ADL). All participants will walk in Alter G one session a day (for 40 min), three days a week, for six weeks. On session one, the Alter G pressure chamber will be set to unload 50% of patient's body weight. On the following sessions, the percentage of unload patient's body weight will be decrease depends on the patient's comfort.
  The physical therapist assistance and treadmill speed will be evaluated and altered based on the patient's capacity. The participants can take a rest whenever his/her need during walking. The rest time will be measured and documented.

SUMMARY:
Stroke is neurological disease characterized by chronic major disability which will cause permanent changes in individuals life. In Saudi Arabia stroke considered as the main leading of disability and death. It is estimated to be 0.67% in Saudi Arabia compared to 2.5% of the population in the United States (US). Most of individuals have mobility deficit such as walk speed and postural maintenance which lead to increase the risk of fall and decrease activity of daily living (ADL).

Stroke rehabilitation should starts as early as possible to avoid post-stroke complications. Several interventions for stroke rehabilitation to improve mobility deficit and posture control continuously being evaluated. One of the ways of stroke rehabilitation is a using of body weight supported treadmill training (BWSTT). It is a useful tool to facilitate gait training and recovery after neurological injures.

The lower body positive pressure (LBPP) is a treadmill that is enclosed in inflated bag. There is a chamber inside the treadmill that is produce air pressure which is aid in eliminate the uncomfortableness feeling produce by weight bearing during gait. The chamber is supplied with a system provide LBPP aiding in decrease patient weight while walking by giving the patient lifting force from below using air pressure. This helps the patient to walk affectively with minimum weight bearing on the lower extremity.

Therefore, the purpose of the study is to evaluate the feasibility and effectiveness of LBPP on gait function, balance and quality of life in chronic stroke individuals.

The investigators hypothesis that the LBPP will significantly improve gait function, balance, quality of life in chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis due to stroke; at least 6 months since the stroke.
* Independent ambulatory ability with or without assistive device at least 10 meters.
* Do not have any additional neurological and/or orthopedic deficiencies impairing ambulation.
* Functional ambulation ≥ 3 on functional ambulation categories
* No history of cardiac, respiratory, cardiovascular conditions interferes with protocol,
* Able to understand simple instructions,
* Able to control the head and trunk posture.

Exclusion Criteria:

* recurrent stroke,
* spasticity greater than 3 on modified Ashowrth scale,
* Ataxia, or tremor of lower limb

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Participation's safety questionnaire as assessed by numerical rating scale rating from 0 (extremely dissatisfied) - 5 (extremely satisfied). | Report the safety at 6 weeks
  The safety of the LBPP will be evaluated by the participation's safety questionnaire. The safety will be measured using numerical rating scale rating from 0 (extremely dissatisfied) - 5 (extremely satisfied). The participant will be asked to rate his/her level of satisfaction for safety variable at the end of 6th weeks.
Participation's satisfaction questionnaire include (comfort, dimensions, personal acceptance, and simplicity of use) will be measured using numerical rating scale rating from 0 (extremely dissatisfied) - 5 (extremely satisfied). | Report the feasibility at 6 weeks
  The feasibility of the LBPP will be evaluated by the participation's satisfaction questionnaire include (comfort, dimensions, personal acceptance, and simplicity of use) will be measured using numerical rating scale rating from 0 (extremely dissatisfied) - 5 (extremely satisfied). The participant will be asked to rate his/her level of satisfaction for each variable at the end of 6th weeks.
Number of participants who have adverse event as assessed by CTCAE v4.0 | Through study completion, an average of 1 year.
  Reporting the presence (or absence) of adverse events
Number of sessions | Through study completion, an average of 1 year.
  Reporting the number of sessions for each participant.
Number of device limitation as assessed by Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) | Through study completion, an average of 1 year.
  Reporting any device limitation that appear during the study

SECONDARY OUTCOMES:
gait function as assessed by 10MWT | Change from baseline gait at 6 weeks.
  10-Meter Walk Test (10MWT): The 10MWT assesses self-selected preferred walking speed over a short duration with or without an assistive device. The participant will be asked to walk a total of 10 meters where an acceleration zone is used for the participants to accelerate 2 meters before entering the 6-meter distance and 2 meters to decelerate afterwards. Speed is only calculated for the 6m distance between the end zones. The 10MWT is widely used in clinical practice and research for people with stroke and has been shown to have an excellent test-retest reliability (ICC > 0.95). The test will be performed three times and the average will be calculated for analysis.
Balance function | Change from baseline balance at 6 weeks.
  Functional Reach Test (FRT): It is used to evaluate participant's stability by measuring the maximum distance participant can reach forward while standing in fixed position. The participant will be standing close to a wall and position the arm at 90 degrees of shoulder flexion close but not touching to the wall with close fist. Starting position will be recorded at the 3rd metacarpal head on yardstick. The participant will be asked to reach as far as he/she can forward with the non-paretic arm without taking a step. The maximum distance that the participant can reach will be recorded. The difference between the start and end position will be calculated. The participant will be allowed for two practice trials. Then, the participant will be asked to perform the test three trials. The average of the three trials will be used for analysis. The FRT showed high intra-rater reliability (ICC = 0.98) and validity (r = 0.71)
Quality of life as assessed by (Short Form 36) | Change from baseline quality of life at 6 weeks.
  Quality of life (Short Form 36): A survey that uses to evaluate quality of life in clinical practice and research purpose. It consist of 8 dimensional subscales: physical functioning, role limitations due to physical problems, general health perceptions, vitality, social functioning, role limitations due to emotional problems, general mental health, and health transition. It has been translated and validated into Arabic language. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. So a high score defines a more favorable health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical City in Qassim University, Buraidah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Almutairi SM, Alfouzan MM, Almutairi TS, Alkaabi HA, AlMulaifi MT, Almutairi MK, Alhuthaifi FK, Swank C. The Safety and Feasibility of Lower Body Positive Pressure Treadmill Training in Individuals with Chronic Stroke: An Exploratory Study. Brain Sci. 2023 Jan 18;13(2):166. doi: 10.3390/brainsci13020166. PMID 36831709